CLINICAL TRIAL: NCT07384039
Title: Effects of Individually Tailored Exercise on Quality of Life and Physical Performance in Patients With Myeloproliferative Neoplasms-a Randomized Controlled Study
Brief Title: Exercise Training in Patients With Myeloproliferative Neoplasms
Acronym: MPN-Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12068-BO-S-2025
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Myeloproliferative Neoplasms (MPN)
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training Group (Experimental): Patients randomized to the 3-month guided exercise training program
  Interventions: Behavioral: Exercise Training
- Wait-List Control Group (No Intervention): Patients randomized to the wait-list control group will maintain their usual lifestyle for the three months intervention period. After this period, they will have the opportunity to participate at the same intervention provided to the exercise training group.

INTERVENTIONS:
Behavioral: Exercise Training — The intervention includes structured and tailored physical training with individual feedback and adjustments to training frequency, intensity, time and content for a total duration of 3 months. Daily activity is monitored using a wearable activity device (Vivoactive 5, Garmin, Olathe, Kansas, USA). An individual training plan includes moderate endurance and strength exercises usually 3 times a week, with the goal of being physically active for at least 150 minutes per week. Participants receive feedback at least every second week via telemonitoring or in person, depending on their distance from the study center. To avoid overexertion, training is monitored by measuring heart rate and providing individual feedback for adjustments if neccesary.
  Arms: Exercise Training Group

SUMMARY:
The investigators will investigate the response of an individualized exercise training program on quality of life, cardiorespiratory fitness and disease-specific markers in patients with myeloproliferative neoplasms (MPN). To this end, the investigators will randomly assign patients with MPN to a training group and a waiting control group.

The training group will undergo an individually tailored exercise training program for three months, while the control group will maintain their usual lifestyle for three months and then has the opportunity to undergo the three-month intervention program. At the beginning and at the end of the three-month intervention phase, the investigators will evaluate physical performance, daily physical activity, muscular strength, and self-reported outcomes and compare them between the training and the control group, in order to assess potential benefits of the exercise training program.

DETAILED DESCRIPTION:
To date, there have been no randomized intervention studies on the effects of physical training in patients with myeloproliferative neoplasms (MPN). Current leukemia and hematology society recommendations and guidelines support the engagement in regular physical activity to improve cardiovascular health, reduce fatigue, and enhance quality of life. However, no disease-specific exercise guidelines for patients with MPNs exist due to the lack of appropriate clinical trials adressing this issue. The aim of the planned study is to investigate an individually tailored physical exercise program with online monitoring for patients with MPN and to measure its effects on quality of life and physical fitness. The primary endpoint is performance (watts) at the respiratory compensation point (RCP), an established marker of submaximal physical performance.

This is a monocentric, prospective, randomized intervention study with a waiting control group. Randomization is performed in a 1:1 ratio to the study groups and is stratified for gender (male/female). The persons conducting the exercise tests (but not the trainers guiding the training program) are blinded so that there is no targeted motivation during the performance test of the intervention group.

Description of the study procedure: The intervention lasts 3 months. The waiting-control group receives the intervention after the 3-month control phase. Participants receive feedback every second week during intervention via telemonitoring or in person, depending on their distance from the study center.

The intervention includes structured, individually tailored physical training with feedback and adjustments to physical activity intensity and content. Daily activity is monitored using a wearable activity device (Garmin smartwatch). An individual training plan includes moderate endurance and strength exercises 3 times a week, with the goal of being physically active for 150 minutes per week. To avoid overexertion, training is monitored by measuring heart rate and providing individual feedback to patients.

The primary evaluation follows the intention-to-treat (ITT) principle, with missing values at the final examination replaced by the corresponding baseline values. An analysis of covariance (ANCOVA) model is used for performance at the RCP, with the mean after-before difference as the primary target variable. Covariates included in the model are the therapy group (intervention and waiting list control), the baseline values of the performance parameter, and gender (female/male). The intervention is considered successful if the lower limit of the two-sided 95% confidence interval is greater than 0.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* diagnosis of myeloproliferative neoplasia according to WHO/ICC 2022.

Exclusion Criteria:

* current participation in another intervention study
* the presence of any diseases or functional impairments that, in the opinion of the examining physician, exclude participation in a physical training intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-04 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in power output (in watt) at the respiratory compensation point (RCP) | From baseline to the end of the intervention period at 3 months
  During an incremental exercise test on a bicycle ergometer power output and gas exchange will be measured continuously. Afterwards the RCP (also known as second ventilatory threshold) will be assessed based on the inflection point of the slopes of the tidal volume (VE) and the carbon dioxide output (VCO2).

SECONDARY OUTCOMES:
Change of the Myeloproliferative Neoplasm-10 (MPN-10) score by 30% (yes/no) | From baseline to the end of the intervention period at 3 months
  Evaluation of the MPN-10, a validated, patient-reported outcome questionnaire specifically designed to assess the symptoms and quality of life in patients with myeloproliferative neoplasms. MPN-10 assesses 10 key symptoms commonly experienced by MPN patients.
  Scoring: 0-4 scale per item, total score ranges from 0 to 40. If the total score is reduced by 30% the binary outcome (yes/no) is fulfilled.
Change in peak oxygen uptake (VO2 in ml/min/kg) | From baseline to the end of the intervention period at 3 months
  During an incremental bicycle exercise test until voluntary exhaustion gas exchange will be measured continuously breath by breath. Within the last stage, the highest oxygen uptake values from single breaths during 30 consecutive seconds are determined as the peak oxygen uptake.
Change in daily physical activity (MET-hours/week) | From baseline to the end of the intervention period at 3 months
  To estimate the total and exercise-related physical activity, metabolic equivalents of task (MET) as MET-hours per week will be calculated, using the International Physical Activity Questionnaire (IPAQ-long) as self-reported outcome
Change in EORTC QLQ-C30 scores | From baseline to the end of the intervention period at 3 months
  The European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 is an internationally used, standardized questionnaire from the European Organization for Research and Treatment of Cancer (EORTC) that assesses health-related quality of life (HrQoL) in cancer patients, measuring functioning (physical, role, emotional, cognitive, social) and symptoms (fatigue, pain, nausea/vomiting). It uses scales from 0-100, where higher scores mean better function/HrQoL (for function scales) or worse symptoms (for symptom scales). Further, a summary score can be calculated by averaging 13 scales (after reversing symptom scales) to provide one overall measure of HrQoL, with higher scores meaning better functioning/HrQoL, and scores range from 0-100.
Change in the FACT-Leu Score | From baseline to the end of the intervention period at 3 months
  The Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) is a valid measure of leukemia-specific health-related quality of life (HrQoL) for acute and chronic disease. Assessed subscales include Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, and a Leukemia Subscale with overall 44 items that has to be responded on a 5 point Likert-type scale. Subscale scores and a total score with a range from 0 to 176 points are possible, with higher scores indicate better HrQoL.

OTHER OUTCOMES:
Change in power output (in watt) at the Ventilatory Threshold (VT) | From baseline to the end of the intervention period at 3 months
  During the incremental exercise test on a bicycle ergometer power output and gas exchange will be measured continuously. Afterwards the VT will be assessed based on the inflection point of the slopes of the carbon dioxide output (VCO2) and the ventilated oxygen (VO2).
Change in steps per day | From baseline to the end of the intervention period at 3 months
  Number of steps will be recorded by a wearable activity tracker (Vivoactive 5, Garmin, Olathe, Kansas, USA) during 7 consecutive days. Valid days will be averaged to get the outcome steps/day.
Change in lactate dehydrogenase (LDH in U/L) | From baseline to the end of the intervention period at 3 months
  LDH is released into the bloodstream upon cellular damage or increased turnover. In patients with MPNs, elevated LDH levels are commonly observed and are associated with increased disease burden, tumor cell proliferation, and adverse prognosis. LDH serves as a non-specific but clinically useful biomarker of disease activity and metabolic stress.
Change in platelet count (in Tsd./µl ) | From baseline to the end of the intervention period at 3 months
  Platelet count is a key component of the complete blood count and reflects bone marrow activity and hemostatic function. In MPNs abnormal platelet production is a hallmark feature, often leading to sustained thrombocytosis (elevated platelet count). Elevated platelet counts are associated with increased risk of thrombotic and hemorrhagic complications, which are major clinical concerns in MPN management.
Change in growth differentiation factor 15 (GDF15 in ng/l) | From baseline to the end of the intervention period at 3 months
  GDF15 is produced by a variety of tissues in response to cellular stress, inflammation, oxidative damage, and mitochondrial dysfunction. Elevated serum GDF15 levels are associated with aging, chronic inflammation, and several hematologic and malignant conditions. In MPNs, GDF15 is often upregulated due to increased bone marrow stress, dysregulated hematopoiesis, and systemic inflammation. Higher GDF15 levels correlate with disease burden, symptom burden, and adverse outcomes, making it a potential biomarker of disease activity and systemic stress.
Change in soluble interleukin-2 receptor (sIL-2R in KU/l) | From baseline to the end of the intervention period at 3 months
  SIL-2R serves as a biomarker of immune system activation and lymphocyte proliferation. Elevated serum levels of sIL-2R are associated with chronic inflammation, autoimmune disorders, and hematologic malignancies. In MPNs, persistent immune dysregulation and chronic inflammation contribute to disease pathogenesis and symptom burden, and sIL-2R levels often correlate with disease activity, inflammatory burden, and clinical progression.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Tegtbur, Prof. Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results of the publication will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 6 months after publication and ending 5 years after publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals should be directed to sportmedizin@mh-hannover.de to gain access, data requestors will need to sign a data-use agreement.